CLINICAL TRIAL: NCT05788224
Title: The Management of Complicated Colo-rectal Cancer in Older Patients in the Emergency Setting: the CO-OLDER Study
Acronym: CO-OLDER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poissy-Saint Germain Hospital (Other)
Collaborators: Fausto Catena (Unknown); World Society of Emergency Surgery (Other)
Responsible Party: Principal Investigator, Belinda De Simone, Principal Investigator, World Society of Emergency Surgery
Other Study IDs: BDS02
Record Dates: First submitted 2023-03-14; First posted 2023-03-28 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Advanced Colorectal Cancer in Elderly Patient
Keywords: elderly; oldest; colorectal cancer; perforation; bleeding; obstruction; emergency; surgery; laparotomy; laparoscopy; futility; frailty
MeSH Terms: conditions — Colorectal Neoplasms; Hemorrhage; Bites and Stings; Emergencies; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter observational study aimed to investigate the management of older patients aged 75 years old and over admitted to the emergency department with complicated colorectal cancer.

The final endpoint is to report morbidity and mortality in this group of frail individuals according to the shift of incidence of colorectal cancer in geriatric patients, over 2 periods: before the COVID pandemic outbreak (11th March 2020) and after the 11th March, during the ongoing pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years old and over;
* Admission to the emergency department with acute abdominal pain;
* Diagnosis of obstructed and/or perforated colorectal cancer.

Exclusion Criteria:

* Patients aged< 75 years old;
* Patients aged >=75 years old admitted with acute abdomen, not due to complicated colorectal cancer.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All older (aged 75 years old and over) patients who were admitted to the surgical department with acute abdominal pain due to a complication of colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
mortality and morbidity correlated with the management of older (=>75 years old) patients admitted to emergency department with a complicated colorectal cancer | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Belinda De Simone, MD, Principal Investigator — World Society of Emergency Surgery
Locations (1):
- World Society of Emergency Surgery, Paris, France

REFERENCES:
- [Derived] DE Simone B, Abu-Zidan FM, Podda M, Pellino G, Sartelli M, Coccolini F, DI Saverio S, Biffl WL, Kaafarani HM, Moore EE, Dhesi JK, Moug S, Ansaloni L, Avenia N, Catena F; CO-OLDER Collaborators. The management of complicated colorectal cancer in older patients in a global perspective after COVID-19: the CO-OLDER WSES project. Minerva Surg. 2024 Jun;79(3):273-285. doi: 10.23736/S2724-5691.23.10165-1. PMID 38847766